CLINICAL TRIAL: NCT01053949
Title: A Multicenter Randomized Open Label Phase II Study of Pomalidomide and Dexamethasone in Relapse and Refractory Multiple Myeloma Patients Who Are Progressive and Did Not Achieve at Least a Partial Response to Bortezomib and Lenalidomide
Brief Title: IFM2009-02-Pomalidomide and Dexamethasone Phase 2 Myeloma
Acronym: IFM2009-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009_28/0924; 2009-013319-36 (EudraCT Number)
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; dexamethasone; pomalidomide; response; safety
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug on 21 days per 28 days cycle (Active Comparator): Pomalidomide 4 mg continuous daily oral route on 21 days per 28 days cycle. The proposed dose of dexamethasone is considered standard, 40mg/day once a week.
  Interventions: Drug: Pomalidomide
- Drug on 28 days per 28 days cycle (Active Comparator): Pomalidomide 4 mg continuous daily oral route on 28 days of a 28 days cycle The proposed dose of dexamethasone is considered standard, 40mg/day once a week.
  Interventions: Drug: Pomalidomide

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide 4 mg continuous daily oral route on 21 days per 28 days cycle. The proposed dose of dexamethasone is considered standard, 40mg/day once a week.
  Other Names: Actimid; CC-4047
  Arms: Drug on 21 days per 28 days cycle
Drug: Pomalidomide — Pomalidomide 4 mg continuous daily oral route on 28 days of a 28 days cycle The proposed dose of dexamethasone is considered standard, 40mg/day once a week.
  Other Names: Actimid; CC-4047
  Arms: Drug on 28 days per 28 days cycle

SUMMARY:
The purpose of this study is to evaluate the response to pomalidomide and dexamethasone in relapse and refractory MM patients who are progressive and did not achieve at least a partial response to bortezomib and lenalidomide. This study will determine the efficacy and toxicity profile of 2 modalities of pomalidomide in patients with advanced myeloma, previously heavily treated characterized with adverse prognostic and that are in desperate need of novel therapeutics.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is an incurable disease that is characterized by the accumulation of clonal plasma cells in the bone marrow. The median overall survival for patients with MM is approximately 4-5 years. Despite front line treatment approaches, the disease eventually relapses. The recent US Food and Drug Administration (FDA) approvals of bortezomib (2003) and combination lenalidomide plus dexamethasone (2006) therapies for the treatment of previously treated MM has provided effective therapeutic options that give patients with relapsed or refractory MM the prospect for a prolongation of overall and progression-free survival times. However, MM remains an incurable disease. A clear unmet medical need still exists for additional novel therapeutic options for the treatment of previously treated MM.

Pomalidomide belongs to the IMiDs class of compounds which thalidomide is the parent compound and lenalidomide the most recently approved agent. It is derived from thalidomide and shares a number of the beneficial pharmacologic properties with thalidomide. The efficacy of thalidomide has been limited by adverse effects. This toxicity profile seems dose and duration-related, spurring the development of IMiDs, which have the potential of improved potency and reduced toxicity. By modifying the thalidomide structure through the addition of an amino group at the 4 position of the phthaloyl ring to generate pomalidomide, a compound that is up to 50000 times more potent at inhibiting TNF-alpha than thalidomide was formed.

Recently, preliminary efficacy and safety data from an ongoing phase 2 study, led by Martha Lacy, et al, at Mayo Clinic, were presented at the XII International Myeloma Workshop in Washington DC (01 March 2009). The study highlighted a 63 % objective response and a 5% complete response in patients taking pomalidomide (2 mg daily on days 1-28 of a 28-day cycle) plus dexamethasone (40 mg daily on days 1, 8, 15, 22 of each cycle) including patients with lenalidomide resistant refractory multiple myeloma. The results also showed that the treatment was well tolerated. Based on the encouraging data of this study, a phase 1/2b multi-center, randomized, open-label, dose escalation study (dose level from 2 mg to 5 mg daily on days 1-21 of a 28-day cycle)is conducted to determine the MTD of pomalidomide. This ongoing study will evaluate the safety and efficacy of oral pomalidomide alone, and in combination with dexamethasone, in patients with relapsed and refractory MM. The first results obtained in this study demonstrated that the maximum tolerated dose of pomalidomide was 4 mg once per day and highlighted that pomalidomide has significant efficacy in MM and can be safely administered to myeloma patients. Moreover, there are an increasing number of patients who are refractory or did not respond significantly or experienced significant toxicity to either bortezomib or lenalidomide.

Based on these studies, we hypothesized that these patients might benefit from the combination of pomalidomide and dexamethasone. We have therefore designed a multicenter phase 2 randomized open labelled study to determine response to pomalidomide and dexamethasone in relapse and refractory MM patients who are progressive and did not achieve at least a partial response to bortezomib and lenalidomide. This study will determine the efficacy and toxicity profile of 2 modalities of pomalidomide in patients with advanced myeloma, previously heavily treated characterized with adverse prognostic and that are in desperate need of novel therapeutics. This study will be conducted in accordance with "good clinical practice" (GCP) and all applicable regulatory requirements, including, where applicable, the 2008 version of the Declaration of Helsinki.

ELIGIBILITY:
Key inclusion criteria:

* Must be able to understand and voluntarily sign an informed consent form
* Must be able to adhere to the study visit schedule and other protocol requirements
* 18 years>=Age
* Life expectancy>6 months
* Patients must have Symptomatic and Progressive Myeloma following bortezomib and/or lenalidomide treatment, defined as detailed in protocol.
* Patients must have a clearly detectable and quantifiable monoclonal M-component value*
* ECOG performance status score of 0,1,or 2
* Adequate bone marrow function,documented within 72 hours prior to treatment without transfusion or growth factor support,defined as*
* Wash out period of at least 2 weeks from previous antitumor therapy or any investigational treatment
* Able to take antithrombotic medicines such as Low molecular weight heparin or Aspirin 75mg
* Subjects affiliated with an appropriate social security system
* Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy
* Agree not to share study medication with another person and to return all unused study drug to the investigator
* Female subjects of childbearing potential* must:Understand that the study medication is expected to have a teratogenic risk-Agree to use,and be able to comply with, effective contraception* without interruption,4 weeks before starting study drug,throughout the entire duration of study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy,even if she has amenorrhoea.This applies unless the subject commits to absolute and continued abstinence on a monthly basis-Understand that even if she has amenorrhea,she must follow all the advice on effective contraception-She understands the potential consequences of pregnancy and the need to rapidly consult if there is a risk of pregnancy-Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/mL on the day of the study visit or in the 3 days prior to the study visit once the subject has been on effective contraception for at least 4 weeks-Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment,except in the case of confirmed tubal sterilization. These pregnancy tests should be performed on the day of the study visit or in the 3 days prior to the study visit.This requirement also applies to women of childbearing potential who practice complete and continued abstinence
* Male subjects must:Agree to use condoms throughout study drug therapy,during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception Agree not to donate semen during study drug therapy and for one week after end of study drug therapy

Exclusion Criteria:

* Any other uncontrolled medical condition or comorbidity that might interfere with subject's participation
* Pregnant or breast feeding females
* Use of any other experimental drug or therapy within 15 days of screening.
* Known positive for HIV or infectious hepatitis,type A, B or C.
* Patients with non-secretory MM
* Prior history of malignancies, other than multiple myeloma, unless the patients has been free of the disease for >= 3 years.Exceptions include the following*
* Prior local irradiation within two weeks before screening
* Evidence of central nervous system involvement
* Any>grade 2 toxicity unresolved
* Peripheral neuropathy>=Grade 2
* Known Hypersensitivity to Thalidomide,Lenalidomide or Dexamethasone
* Ongoing active infection,especially ongoing pneumonitis
* Ongoing Cardiac dysfunction
* Inability or unwillingness to comply with birth control requirements
* Unable to take antithrombotic medicines at study entry
* Unable to take corticotherapy at study entry
* Refusal to participate in the study
* Persons protected by a legal regime(guardianship,trusteeship)

(*)=described in protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-10; Primary Completion 2014-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
To determine Response rate to pomalidomide and dexamethasone in MM patients who are progressive and did not achieve at least a partial response to bortezomib and lenalidomide | 30 months

SECONDARY OUTCOMES:
To determine response and safety profile of 2 dose-regimens of pomalidomide | 30 months
To determine Safety of pomalidomide and dexamethasone | 30 months
To determine Time to response and Response duration of pomalidomide and dexamethasone | 30 months
To determine Time to disease progression to pomalidomide and dexamethasone | 30 months
Overall Survival of pomalidomide and dexamethasone | 30 months
To determine response in both arms with regards to cytogenetic of the bone marrow tumor plasma cells | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno ROYER, MD PhD, Principal Investigator — CHRU-Hôpital Sud d'Amiens-AMIENS; Philippe RODON, MD PhD, Principal Investigator — Centre Hospitalier de Blois -BLOIS; Sabine BRECHIGNAC, MD PhD, Principal Investigator — Hôpital Avicenne-Bobigny- PARIS; Gerard MARIT, MD PhD, Principal Investigator — Hôpital Haut-Levèque de Pessac-BORDEAUX; Christian BERTHOU, MD PhD, Principal Investigator — Service d'Hématologie Clinique, CHU Morvan, BREST; Margaret MACRO, MD PhD, Principal Investigator — Hématologie, CHU, CAEN; Denis CAILLOT, MD PhD, Principal Investigator — Hématologie Clinique, CHU, Hôpital d'Enfants, DIJON; Brigitte PEGOURIE, MD PhD, Principal Investigator — Hématologie, CHRU, Hôpital A.Michallon, GRENOBLE; Catherine TRAULLE, MD PhD, Principal Investigator — Service d'Hématologie, Centre Hospitalier Lyon Sud, PIERRE BENIT; Anne Marie STOPPA, MD PhD, Principal Investigator — Hématologie, Institut Paoli Calmette, MARSEILLE; Cyrille HULIN, MD PhD, Principal Investigator — Hématologie, CHRU, Hôpitaux de Brabois, VANDOEUVRE; Philippe MOREAU, MD PhD, Principal Investigator — Maladies du Sang, CHRU, Hôtel Dieu, NANTES; Jean-Gabriel FUZIBET, MD PhD, Principal Investigator — Médecine Interne, Oncologie, Hôpital de l'Archet 1, NICE; Bernard GROSBOIS, MD PhD, Principal Investigator — Médecine Interne, CHRU, Hôpital Sud, RENNES; Brigitte KOLB, MD PfD, Principal Investigator — Hématologie Clinique, Hôpital Robert Debré, CHU REIMS; Laurent GARDERET, MD PhD, Principal Investigator — Maladies du Sang, CHU - Hôpital St Antoine, PARIS; Jean-Paul FERMAND, MD PhD, Principal Investigator — Service Immuno-Hématologie, Hôpital Saint-Louis, PARIS; Michel ATTAL, MD PhD, Principal Investigator — Hématologie, CHRU, Hôpital Purpan, TOULOUSE; Lofti BENBOUBKER, MD PhD, Principal Investigator — Onco-Hématologie, CHRU- Hôpital Bretonneau, TOURS; Xavier Leleu, MD PhD, Study Director — Service des maladies du sang, CHRU de Lille
Locations (19):
- France (19):
  - CHRU-Hôpital Sud, avenue Laennec,, Amiens
  - Hématologie, Hôpital Avicenne, Bobigny
  - Hématologie, CHU, avenue G.Clemenceau, Caen
  - Hématologie Clinique, CHU, Hôpital d'Enfants, Dijon
  - Hématologie, CHRU, Hôpital A.Michallon, Grenoble
  - Service des Maladies du Sang, CHRU, Lille
  - Hôpital Edouard HERRIOT, Lyon
  - Hématologie, Institut Paoli Calmette, Marseille
  - Hématologie, CHRU, Hôpitaux de Brabois, Nancy
  - Maladies du Sang, CHRU, Hôtel Dieu, Nantes
  - Service Immuno-Hématologie, Hôpital Saint-Louis, Paris
  - Maladies du Sang, CHU - Hôpital St Antoine, Paris
  - Service des Maladies du Sang, Hôpital Haut-Levèque, Pessac
  - Service d'Hématologie, Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hématologie Clinique, Hôpital Robert Debré, CHU Reims, Reims
  - Hôpital PONTCHAILLOU, CHU de RENNES, Rennes
  - Médecine Interne, CHRU, Hôpital Sud, Rennes
  - Hématologie, CHRU, Hôpital Purpan, Toulouse
  - Onco-Hématologie, CHRU- Hôpital Bretonneau, Tours

REFERENCES:
- [Derived] Leleu X, Attal M, Arnulf B, Moreau P, Traulle C, Marit G, Mathiot C, Petillon MO, Macro M, Roussel M, Pegourie B, Kolb B, Stoppa AM, Hennache B, Brechignac S, Meuleman N, Thielemans B, Garderet L, Royer B, Hulin C, Benboubker L, Decaux O, Escoffre-Barbe M, Michallet M, Caillot D, Fermand JP, Avet-Loiseau H, Facon T; Intergroupe Francophone du Myelome. Pomalidomide plus low-dose dexamethasone is active and well tolerated in bortezomib and lenalidomide-refractory multiple myeloma: Intergroupe Francophone du Myelome 2009-02. Blood. 2013 Mar 14;121(11):1968-75. doi: 10.1182/blood-2012-09-452375. Epub 2013 Jan 14. PMID 23319574